CLINICAL TRIAL: NCT05573022
Title: Impact of a Patient Decision Aid Intervention for Cancer Patients. Does Timing and Format Matter?
Brief Title: Impact of a Patient Decision Aid Intervention
Acronym: IMPACTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: The Ottawa Hospital Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMPACTT
Record Dates: First submitted 2022-09-20; First posted 2022-10-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cancer, Breast; Cancer Colorectal
Keywords: Shared decision making; Patient decision aids; Patient preferences; Patient engagement
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Patient Preference; Patient Participation

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomised, controlled trial, in which patients are allocated to either a digital pre-consultation patient decision aid or a paper-based in-consultation patient decision aid. A total estimate of 204 patients with breast and 70 patients with colorectal cancer are included in the study including 10% to compensate for missing data and dropouts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A1: Breast cancer patients (Experimental)
  Interventions: Other: Pre-consultation electronic patient decision aid
- Arm B1: Breast cancer patients (Active Comparator)
  Interventions: Other: In-consultation paper-based patient decision aid
- Arm A2: Colorectal cancer patients (Experimental)
  Interventions: Other: Pre-consultation electronic patient decision aid
- Arm B2: Colorectal cancer patients (Active Comparator)
  Interventions: Other: In-consultation paper-based patient decision aid

INTERVENTIONS:
Other: Pre-consultation electronic patient decision aid — This group is invited to access an electronic version before the consultation. The group of colorectal cancer patients is also introduced to a paper-based version by the clinician in the consultation.
  Arms: Arm A1: Breast cancer patients; Arm A2: Colorectal cancer patients
Other: In-consultation paper-based patient decision aid — This group is introduced to a paper-based version by the clinician in the consultation
  Arms: Arm B1: Breast cancer patients; Arm B2: Colorectal cancer patients

SUMMARY:
Studies evaluating decisions aids have used a wide range of outcome measures as well as formats and settings. Most studies have focused on patient decision aids used either within the consultation or delivered pre-consultation, but there are no randomised, controlled studies comparing the two. However, timing and format of the patient decision aid intervention may affect how useful the tool is to the patient. The aim of this project is therefore to deepen our understanding of the patient's engagement in and preparation for the decision making process in a randomised, controlled trial comparing an electronic pre-consultation and paper-based in-consultation patient decision aid. 274 patients with colorectal and breast cancer are enrolled in the study. Data are collected at both patient and consultant perceived levels as well as an observed level of shared decision making.

DETAILED DESCRIPTION:
A cancer diagnosis is life-changing and followed by complex decisions about treatment options. Often the decision about which treatment to choose is based on risks and benefits, although the benefit-harm ratios are unknown. In these situations, a patient decision aid can be helpful in explaining the options, clarifying the patient's preferences and acting as an adjunct to the clinician's counselling, supporting the patient in complex decisions about their diagnosis.

Studies evaluating patient decision aids have used a wide range of outcome measures as well as formats and settings. Most studies have focused on patient decision aids used either within the consultation or delivered pre-consultation, but there are no randomised, controlled studies comparing the two. There is a lack of evidence of the impact of patient decison aids used pre-consultation versus in-consultation, as timing and format of the patient decision aid intervention may affect how useful the tool is to the patient. The aim of this project is therefore to deepen our understanding of the patient's engagement in and preparation for the decision making process in a randomised, controlled trial comparing a digital pre-consultation and paper-based in-consultation patient decision aid. 274 patients with colorectal and breast cancer are enrolled in the study. Data are collected at both patient and consultant perceived level as well as an observed level of shared decision making (SDM).

A secondary analysis of the data collected in the study will form the basis of a study testing the convergent validity of the patient-reported measures by comparing them to the observed level of patient involvement. During the last decade, the strong move towards increased SDM has led to development of several measurement scales, and there is a demand for convergent validity studies, as there is no gold standard to evaluate SDM behaviors. Previous validity studies have various shortcomings.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified breast or colorectal cancer
* Age ≥ 18 years

Exclusion Criteria:

* Unable to read Danish
* Not the owner/user of a mobile smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Level of involvement of patients in shared decision making (breast cancer) | Within one week after the consultation
  4-item Shared Decision Making Process Scale (SDM Process 4) with patient-reported measures of the amount of shared decision making that occurs around the medical decision. Score range is 0 to 4 points, a higher score indicates more involvement in the decision.
Observed level of patient involvement in decision making according to the OPTION5 tool (colorectal cancer) | Through study completion, an average of 3 months
  settings (OPTION5). Scores range 0-100. Higher score indicates higher patient involvement in decision making.

SECONDARY OUTCOMES:
Patient-perceived level of shared decision making (breast and colorectal cancer) | Within one week after the consultation
  9-item Shared Decision Making Questionnaire (SDM-Q-9) that measures the extent to which patients are involved in the process of decision-making from the perspective of the patient. Scores range from 1 to 6 on each question. The total score range is thus 9-54 with 54 as the best score indicating higher involvement.
Patient-perceived level of shared decision making between patient and consultant (breast and colorectal cancer) | Within one week after the consultation
  3-item questionnaire (CollaboRATE) with patient-reported measures of the perception of being informed and involved in decision making. Each item is scored on a 0 to 9 scale on a 10-point Likert scale, a higher score indicates a better experience.
Level of patient preparation for decision making (breast and colorectal cancer) | Within one week after the consultation
  10-item questionnaire (Preparation for Decision Making Scale) with patient-reported measures of how useful the decision aid / decision support intervention is in preparing the patient for the consultation. The scale is from 1 (not at all useful) to 5 (very useful). Higher scores indicate greater preparation.
Level of decisional conflict (breast and colorectal cancer) | Before consultation and within one week after the consultation
  16-item questionnaire (Decisional conflict scale) with patient-reported measures of uncertainty and decisional conflict. Each item is rated on a 5-point scale, and total scores are calculated by summing the raw scores of all items and presenting them on a scale of 0-100, with higher scores indicating greater decision conflict. Scores greater than 25 indicate clinically important decisional conflict.
Degree of control over the decision about medical treatment (breast and colorectal cancer) | Before the consultation
  1-item questionnaire (Control Preference Scale) with a patient-reported measure of the degree of control that the patient wants to assume when decisions are being made about medical treatment. Answers range from Fully active role, Semiactive role, Collaborative role, Semipassive role and Fully passive role.
Consultant-perceived level of shared decision making (breast and colorectal cancer) | Within one week after the consultation
  9-item Shared Decision Making Questionnaire (SDM-Q-doc) that measures the extent to which patients are involved in the process of decision-making from the perspective of the consultant. The items are scored from 0 to 5 on a six-point Likert scale ranging from "completely disagree" (0) to "completely agree" (5). A linear transformation of item score sum yields a transformed score (0-100), with higher values indicating more shared decision making.
Observed level of patient involvement in decision making according to the OPTION5 tool (breast cancer) | Through study completion, an average of 3 months
  Measuring shared decision making by assessing recordings of encounters from clinical settings (OPTION5). Scores range 0-100. Higher score indicates higher patient involvement in decision making.
Level of involvement of patients in shared decision making (colorectal cancer) | Within one week after the consultation
  4-item Shared Decision Making Process Scale (SDM Process 4) with patient-reported measures of the amount of shared decision making that occurs around the medical decision. Score range is 0 to 4 points, a higher score indicates more involvement in the decision.

OTHER OUTCOMES:
Consultation length measured in minutes | Through study completion, an average of 3 months
  Length of consultation in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Karina Dahl Steffensen, Study Chair — Sygehus Lillebaelt
Locations (1):
- Lillebaelt Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make data available to others

REFERENCES:
- [Derived] Knudsen BM, Sondergaard SR, Stacey D, Steffensen KD. Impact of timing and format of patient decision aids for breast cancer patients on their involvement in and preparedness for decision making - the IMPACTT randomised controlled trial protocol. BMC Cancer. 2024 Mar 12;24(1):336. doi: 10.1186/s12885-024-12086-z. PMID 38475758